CLINICAL TRIAL: NCT01718912
Title: The Effect of an Antibiotic-antifungal Rinse on Periodontal Disease
Brief Title: Periodontal Disease Treatment of a Physically Challenged Population
Acronym: PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oravital Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OVTRI; TRI (Other: Toronto Rehabilitation Institute)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Periodontal Disease
Keywords: periodontal disease; bleeding on probing; periodontal pockets; disabled
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metronidazole-nystatin oral rinse, regular oral hygiene (Other): Week 1: daily brushing with suction brush. Week two: daily brushing with a mixture of metronidazole-nystatin suspension.
  Interventions: Drug: metronidazole-nystatin oral rinse

INTERVENTIONS:
Drug: metronidazole-nystatin oral rinse

SUMMARY:
Many physically handicapped patients at the dental department, Toronto Rehabilitation Institute(TRI) have considerable gingival inflammation and breath odour because of the inability to effectively handle a toothbrush. These patients have considerable periodontal disease. There is a concern that these pathogens may have a detrimental effect on wound healing in other areas of the body.

Hypothesis: Patients attending the dental department at TRI that are treated with the antibiotic-antifungal rinse containing metronidazole and nystatin will show substantial decrease in periodontal disease as measured by bleeding points and pocket depth when compared to the group that continues to use their regular oral hygiene methods (control group).

ELIGIBILITY:
Inclusion Criteria:

Participants must be between the ages of 18 to 65 years Participants must have at least 6 teeth. Participants must have some indication of gingivitis and periodontal breakdown. -

Exclusion Criteria:

Patients who are taking Warfarin/Coumadin Patients who are allergic to Metronidazole or chlorhexidine. Edentulous patients will be excluded by those who have at least 6 teeth can be a participant

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evidence of healing of periodontal tissues as shown by a reduction of bleeding | two weeks
  Evidence of healing of periodontal tissues is assessed by measuring bleeding points and periodontal pocket depth using a dental probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Rehabilitation Institute, Dental Department, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No